CLINICAL TRIAL: NCT01059578
Title: A Single Blind, Randomised, Placebo Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GSK206136 in Healthy Male Subjects and an Open Label Positron Emission Tomography Study to Evaluate the Serotonin Transporter and Neurokinin-1 Receptor Occupancy
Brief Title: First Study in Humans With GSK206136
Acronym: NSB101909
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 101909
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Depressive Disorder and Anxiety Disorders
Keywords: Nk1 Antagonist and SSRI; Safety; First Time in Humans; Healthy Subjects
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): GSK206136 once daily
  Interventions: Drug: GSK206136; Radiation: PET
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: GSK206136 — GSK206136 2mg, 10mg, 50mg, 100mg capsule
  Arms: Active
Drug: PLACEBO — Placebo to match 206136 2mg, 10mg, 50mg, 100mg capsule
  Arms: Placebo
Radiation: PET — Each subject will undergo 3 PET Scans ; one at Baseline and the others following dosing with GSK206136 at approximately 2 hours post-dose and 24 hours post-dose
  Arms: Active

SUMMARY:
This is the first study in humans with GSK206136 to evaluate what effects: good or bad, the drug has on human health (safety and tolerability) and the amount of drug which gets into the bloodstream and is eliminated from the body (pharmacokinetics). Also the study aims to investigate the penetration of the drug in the human brain by using PET (Positron Emission Tomography) imaging technology

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 18-45 years, limited to 25-40 years of age for PET section

Exclusion Criteria:

* The subject has a positive: drug/alcohol, Hepatitis, HIV screen..
* The subject has a history of psychiatric illness suicidal attempts or behaviour.
* Abuse of alcohol.
* Clinically significant laboratory, ECG abnormality;
* The subject has recently received an investigational.
* Use of prescription or non-prescription drugs,
* History or presence of allergy to the study drug or drugs of this class,
* Donation of more than 500 mL blood within the 90 days before dosing.
* An unwillingness of male subjects to comply with contraceptive requirements
* Average daily caffeine intake exceeding Protocol requirements.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2006-05-23 (Actual); Primary Completion 2006-12-18 (Actual); Study Completion 2006-12-18 (Actual)

PRIMARY OUTCOMES:
Adverse event monitoring, vital signs (blood pressure, heart rate, ECGs, clinical laboratory assessments (standard laboratory parameters); pharmacokinetics parameters: AUC, Cmax, t1/2 | 12 weeks

SECONDARY OUTCOMES:
Brain receptor occupancy | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- See also: Results for study 101909 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/101909?search=study&search_terms=101909#rs